CLINICAL TRIAL: NCT03004261
Title: Cytomegalovirus Specific Cytotoxic T Lymphocyte for the Treatment of Cytomegalovirus Infection After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: CMV-CTL for the Treatment of CMV Infection After HSCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Principal Investigator, Liping Wan, Chief Physician, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMV-CTL-201609
Record Dates: First submitted 2016-12-18; First posted 2016-12-28 (Estimated); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cytomegalovirus Infections; Hematological Disease
Keywords: cytomegalovirus infection; cytotoxic T lymphocyte; hematopoietic stem cell transplantation
MeSH Terms: conditions — Cytomegalovirus Infections; Hematologic Diseases | interventions — Foscarnet; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CMV-CTL (Experimental): The donor derived cytomegalovirus specific T lymphocytes (CMV-CTL) will be transfused to the patients. The patients will receive CMV-CTL cells when they are sero-positive for CMV-DNA 30 days after transplant. The CMV-DNA levels will be monitored weekly for at least 60 days after the transplant. If after the initial dose of CMV-CTL cells the patient develops a viral infection, then they may be eligible to receive one additional injection of CMV-CTLs. If the CMV levels in the blood continue to rise after the dose of T cells then the patient will receive treatment with Ganciclovir or Foscarnet.
  Interventions: Biological: donor derived cytomegalovirus specific T lymphocytes; Drug: Foscarnet; Drug: Ganciclovir

INTERVENTIONS:
Biological: donor derived cytomegalovirus specific T lymphocytes — donor derived cytomegalovirus specific T lymphocytes will be transfused to recipients of hematopoietic stem cell transplant when they are sero-positive for CMV-DNA.
  Other Names: cytomegalovirus specific T lymphocytes
Drug: Foscarnet — Foscarnet may be used for the treatment of CMV infection before and after the CMV-CTL infusion.
Drug: Ganciclovir — Ganciclovir may be used for the treatment of CMV infection before and after CMV-CTL infusion.

SUMMARY:
Human cytomegalovirus (CMV) infection is a major cause of morbidity and mortality for recipients of allogeneic hematopoietic stem cell transplantation(HSCT). we propose to study the immunologic and virologic effects of donor derived CMV specific cytotoxic T lymphocyte (CMV-CTL) given to transplant recipients

CMV antigen peptides will be used to induce the CMV antigen specific T lymphocytes derived from donor peripheral blood mononuclear cells for a period of 18~21 days.The patients will receive CMV-CTL cells when they are sero-positive for CMV-DNA 30 days after transplant. The CMV-DNA level will be monitored weekly after transfusion.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation is widely used for the treatment of hematological malignancies and bone marrow failure diseases. Human cytomegalovirus (CMV) infection is a major cause of morbidity and mortality for recipients of allogeneic hematopoietic stem cell transplantation(HSCT). Approximately half of the recipients would develop CMV infection after transplant. Present treatment recommendation for CMV infection including ganciclovir and foscarnet. However, these medications have many side effects, the most serious is myelosuppression and renal injury, moreover, many patients do not response to these medications. Considering the risk associated with persistent infection and the potential for CMV specific cytotoxic T lymphocyte (CMV-CTL) to restore immunity, we propose to study the immunologic and virologic effects of donor derived CMV-CTL given to transplant recipients, levels of CMV-CTL and CMV DNA will be measured from CTL recipients.

If the patient and their donor are eligible, we will take 80 ml of fresh blood from the donor or 5 ml peripheral blood stem cell from the donor.The peripheral blood mononuclear cells will be separated from peripheral blood or peripheral blood stem cell. CMV antigen peptides will be used to induce the CMV-CTL for a period of 18~21 days.

The donor derived CMV-CTL cells will be transfused into the patients' intravenous line. The patients will receive the dose of CMV-CTL cells when they are sero-positive for CMV-DNA 30 days after transplant. The CMV-DNA levels will be monitored weekly for at least 60 days after the transplant. If after the initial dose of CMV-CTL cells the patient develops a viral infection, then they may be eligible to receive one additional injection of CTLs. If the CMV levels in the blood continue to rise after the dose of T cells then the patient will receive treatment with Ganciclovir, Foscarnet.

ELIGIBILITY:
Inclusion Criteria:

* Any allogeneic stem cell transplant recipient ≥ 14 years of age and ≤ 60 years of age
* Bilirubin/ SGOT/SGPT < 5 × upper normal limits.
* Creatinine < 2 × upper normal limits.
* Ejection fraction ≥ 50%, no severe arrhythmia.
* Estimated life expectancy ≥ 6 months.
* Patients' CMV-DNA ≥ 1000cp/ml in treatment group and being negative in prophylactic group.

Exclusion Criteria:

* Patients receiving prednisone ≥ 1mg/kg/d for the treatment of acute GVHD or mild, severe chronic GVHD.
* Recipient < 14years of age
* Donor is sero-positive in HBV/HCV/HIV or RPR.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2016-11; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
30-day response rate | from the date of CMV-CTL infusion to 30 days after the infusion
  The percentage of patient whose serum CMV-DNA becomes negative in 30 days.

SECONDARY OUTCOMES:
1-year overall survival | from the date of transplant to 1 year after transplant
  The length of patients who are alive in 1 years.
100-day incidence of acute GVHD | from the date of transplant to 100 days after transplant
  the incidence of acute GVHD
1-year incidence of chronic GVHD | from the date of transplant to 1 year after transplant
  the incidence of chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Liping Wan, M.D.，Ph.D., Principal Investigator — Shanghai Jiao Tong University Affiliated Shanghai General Hospital
Locations (1):
- Shanghai Jiao Tong University Affilated Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No